CLINICAL TRIAL: NCT05342636
Title: A Phase 1/2 Open-Label, Umbrella Platform Design Study of Investigational Agents With or Without Pembrolizumab (MK-3475) and/or Chemotherapy in Participants With Advanced Esophageal Cancer naïve to PD-1/PD-L1 Treatment (KEYMAKER-U06): Substudy 06A.
Brief Title: A Study of Combination Therapies With or Without Pembrolizumab (MK-3475) and/or Chemotherapy in Participants With Advanced Esophageal Cancer (MK-3475-06A)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-06A; 2031220197 (Registry Identifier: JRCT); 2023-505188-36-00 (Registry Identifier: EU CT); U1111-1291-1899 (Registry Identifier: UTN); 2021-005405-26 (EudraCT Number)
Record Dates: First submitted 2022-04-19; First posted 2022-04-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: Esophageal cancer; Programmed Cell Death 1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL-1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL-2, PD-L2)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib; Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pembrolizumab plus chemotherapy (Experimental): Participants will receive pembrolizumab intravenously plus chemotherapy (investigator's choice of irinotecan or paclitaxel) at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Drug: Irinotecan; Drug: Paclitaxel
- Coformulation Favezelimab/Pembrolizumab plus Chemotherapy (Experimental): Participants will receive coformulation of favezelimab/pembrolizumab administered intravenously plus chemotherapy (investigator's choice of irinotecan or paclitaxel) at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Coformulation favezelimab/pembrolizumab; Drug: Irinotecan; Drug: Paclitaxel
- Pembrolizumab plus MK-4830 plus Chemotherapy (Experimental): Participants will receive pembrolizumab intravenously plus MK-4830 plus chemotherapy (investigator's choice of irinotecan or paclitaxel) at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Biological: MK-4830; Drug: Irinotecan; Drug: Paclitaxel
- Pembrolizumab plus MK-4830 plus lenvatinib (Experimental): Participants will receive pembrolizumab intravenously plus MK-4830 plus lenvatinib orally at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Biological: MK-4830; Drug: Lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg administered via intravenous (IV) infusion every 3 weeks (Q3W)
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab plus MK-4830 plus Chemotherapy; Pembrolizumab plus MK-4830 plus lenvatinib; Pembrolizumab plus chemotherapy
Biological: Coformulation favezelimab/pembrolizumab — 800 mg favezelimab + 200 mg pembrolizumab administered via IV infusion on day 1 and then Q3W
  Other Names: MK-4280A
  Arms: Coformulation Favezelimab/Pembrolizumab plus Chemotherapy
Biological: MK-4830 — 800 mg administered via IV infusion Q3W
  Other Names: anti-immunoglobulin-like transcript 4 (ILT4)
  Arms: Pembrolizumab plus MK-4830 plus Chemotherapy; Pembrolizumab plus MK-4830 plus lenvatinib
Drug: Lenvatinib — 20 mg administered via oral capsules each day
  Other Names: MK-7902; LENVIMA®
  Arms: Pembrolizumab plus MK-4830 plus lenvatinib
Drug: Irinotecan — 180 mg/m^2 administered via IV infusion on day 1 of every 14-day cycle.
  Arms: Coformulation Favezelimab/Pembrolizumab plus Chemotherapy; Pembrolizumab plus MK-4830 plus Chemotherapy; Pembrolizumab plus chemotherapy
Drug: Paclitaxel — 80-100 mg/m^2 administered via IV infusion on Days 1, 8 and 15 of every 28 day cycle
  Arms: Coformulation Favezelimab/Pembrolizumab plus Chemotherapy; Pembrolizumab plus MK-4830 plus Chemotherapy; Pembrolizumab plus chemotherapy

SUMMARY:
This is a phase I/II multicenter, open-label umbrella platform study that will evaluate the safety and efficacy of investigational agents with pembrolizumab, plus chemotherapy or lenvatinib, for the treatment of participants with advanced esophageal cancer who have failed 1 prior line of therapy and have not been previously exposed to programmed cell death 1 protein (PD-1)/ programmed cell death ligand 1 (PD-L1) based treatment.

With protocol amendment 5 (effective: 17-November-2023), enrollment in study arms "Pembrolizumab plus MK-4830 plus Chemotherapy" and "Pembrolizumab plus MK-4830 plus lenvatinib" is discontinued.

DETAILED DESCRIPTION:
The master protocol is MK-3475-U06.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic or locally advanced unresectable ESCC
* Has experienced investigator documented radiographic or clinical disease progression on one prior line of standard therapy.
* Has an evaluable baseline tumor sample (newly obtained or archival) for analysis
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications
* Participants who have adverse events (AEs) due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible

Exclusion Criteria:

* Direct invasion into adjacent organs such as the aorta or trachea
* Has experienced weight loss >10% over approximately 2 months prior to first dose of study therapy
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Known additional malignancy that is progressing or has required active treatment within the past 3 years, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that has undergone potentially curative therapy
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in past 2 years
* History of human immunodeficiency virus (HIV) infection
* History of Hepatitis B or known active Hepatitis C virus infection
* History of allogenic tissue/solid organ transplant
* Clinically significant cardiovascular disease within 12 months from first dose of study intervention
* Participants with known gastrointestinal (GI) malabsorption or any other condition that may affect the absorption of lenvatinib
* Has risk for significant GI bleeding, such as:
* Has had a serious nonhealing wound, peptic ulcer, or bone fracture within 28 days prior to allocation/randomization
* Has significant bleeding disorders, vasculitis, or has had a significant bleeding episode from the GI tract within 12 weeks prior to allocation/randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing a Dose-limiting Toxicity (DLT) During Safety Lead-in Phase | Up to approximately 3 weeks
  A DLT is defined as any drug-related adverse event (AE) according to the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) Version 5.0, observed during the DLT evaluation period that results in a change to a given dose or a delay in initiating the next cycle.
Number of Participants Experiencing an Adverse Event (AE) During Safety Lead-in Phase | Up to approximately 3 Weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE During Safety Lead-in Phase | Up to approximately 3 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Objective Response Rate (ORR) | Up to approximately 40 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 40 months
  PFS is defined as the time from allocation to the first documented progressive disease (PD) as assessed by RECIST 1.1 or death due to any cause, whichever occurs first. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Duration of Response (DOR) | Up to approximately 40 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 40 months
  OS is defined as the time from the date of allocation to death from any cause.
Number of Participants Experiencing at Least One Adverse Event (AE) During the Efficacy Phase | Up to approximately 40 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Treatment Due to An AE During the Efficacy Phase | Up to approximately 104 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (46):
- Brazil (3):
  - Liga Norte Riograndense Contra o Câncer ( Site 2303), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceição ( Site 2301), Porto Alegre, Rio Grande do Sul
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO ( Site 2300), São Paulo, São Paulo
- Chile (2):
  - FALP-UIDO ( Site 2400), Santiago, Region M. de Santiago
  - Clínica las Condes ( Site 2403), Santiago, Region M. de Santiago
- France (3):
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital Morvan ( Site 1104), Brest, Finistere
  - Hopital Claude Huriez - CHU de Lille ( Site 1100), Lille, Nord
  - Pitie Salpetriere University Hospital ( Site 1102), Paris, Orne
- Germany (4):
  - Institut für Klinisch Onkologische Forschung-Klink für Onkologie und Hämatologie ( Site 2801), Frankfurt am Main, Hesse
  - Universitaetsklinikum Duesseldorf ( Site 2802), Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Medical Dept I - Medical Oncology ( Site 2806), Dresden, Saxony
  - Charité Campus Virchow-Klinikum-Klinik Hämatologie Onkologie Tumorimmunologie ( Site 2804), Berlin
- Italy (4):
  - Ospedale San Raffaele-Oncologia Medica ( Site 1206), Milan, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1200), Milan, Lombardy
  - Istituto Europeo di Oncologia IRCCS-Divisione di Sviluppo di Nuovi Farmaci per Terapie Innovative (, Milan
  - Istituto Oncologico Veneto IRCCS ( Site 1205), Padua
- Japan (5):
  - Aichi Cancer Center Hospital ( Site 1702), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 1701), Kashiwa, Chiba
  - Saitama Prefectural Cancer Center ( Site 1703), Ina-machi, Saitama
  - Shizuoka Cancer Center ( Site 1704), Nagaizumi-cho,Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 1700), Chuo-ku, Tokyo
- Oslo universitetssykehus, Radiumhospitalet ( Site 2501), Oslo, Norway
- National University Hospital ( Site 1800), Singapore, South West, Singapore
- South Korea (2):
  - Asan Medical Center-Department of Oncology ( Site 1901), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 1900), Seoul
- Switzerland (2):
  - Hôpitaux Universitaires de Genève (HUG) ( Site 2702), Geneva, Canton of Geneva
  - Kantonsspital Graubünden-Medizin ( Site 2700), Chur, Kanton Graubünden
- Taiwan (7):
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 2003), Kaohsiung Niao Sung Dist, Kaohsiung
  - China Medical University Hospital ( Site 2007), Taichung
  - Taichung Veterans General Hospital-Radiation Oncology ( Site 2008), Taichung
  - National Cheng Kung University Hospital ( Site 2001), Tainan
  - National Taiwan University Hospital ( Site 2000), Taipei
  - Taipei Veterans General Hospital ( Site 2005), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 2006), Taoyuan District
- Thailand (3):
  - Chulalongkorn University ( Site 2104), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 2102), Bangkok, Bangkok
  - Songklanagarind hospital ( Site 2105), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (9):
  - Acibadem Altunizade Hospital-Oncology ( Site 1407), Üsküdar / İstanbul, Istanbul
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 1406), Izmir, Karsiyaka, İzmir
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 1417), Adana
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 1402), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 1408), Ankara
  - Ankara City Hospital-Medical Oncology ( Site 1405), Ankara
  - Akdeniz Universitesi Hastanesi-Medical Oncology ( Site 1410), Antalya
  - Atatürk Üniversitesi-onkoloji ( Site 1416), Erzurum
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1403), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26342&tenant=MT_MSD_9011